CLINICAL TRIAL: NCT03618017
Title: Patient-Centered, Team-Based Continuing Care After Breast Cancer Treatment: The ConnectedCancerCare Pilot Study
Brief Title: The ConnectedCancerCare Pilot Study (CCC)
Acronym: CCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UMCC 2018.016; K07CA201052 (NIH); HUM00115786 (Other: University of Michigan)
Record Dates: First submitted 2018-07-13; First posted 2018-08-07 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Early-stage Breast Cancer; Breast Cancer Female; Survivorship; Cancer Survivors; Transitional Care
Keywords: Breast cancer; Survivors; Survivorship plan; Transitional cancer care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized control pilot trial of a web-based, personalized navigation tool to support the continuing and team-based care of early-stage breast cancer patients who have completed their primary cancer treatment. Patients will be randomized to either the intervention (n=30), a personalized website that guides team-based, survivorship care or to the control (n=30), an static online survivorship care plan.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to the intervention (website) or control (informational template) after completing an online questionnaire; they will not be informed of which arm of the study they are participating. The allocation of participants will be masked for the investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCC Website (Experimental): The intervention, ConnectedCancerCare (CCC) Website is a personalized, navigation tool that is tailored to patients' preferences for provider roles in follow-up care, their satisfaction with their current primary care provider, and their worry about cancer recurrence. It involves a personalized, patient-facing website which includes a baseline survey, tailored educational modules, and a guide for their survivorship care, as well as a text or email based reminder system. The intervention also includes a provider-facing summary document, which will be faxed to both the oncology and primary care teams.
  Interventions: Behavioral: CCC website
- Static care plan (Other): The control arm will receive is a static survivorship care plan template in PDF format that includes information similar to what an oncologist currently provides as "standard of care."
  Interventions: Behavioral: Static care plan

INTERVENTIONS:
Behavioral: CCC website — ConnectedCancerCare (CCC) is a web-based guide to support survivorship care for women who have been treated for early-stage (stages 0-II) breast cancer. It encourages patients to utilize team-based care by oncologists and primary care physicians and provides them with the information on cancer surveillance, screenings and preventive healthcare during survivorship.
  Other Names: ConnectedCancerCare
  Arms: CCC Website
Behavioral: Static care plan — The control is a static survivorship care plan template in PDF format that includes information similar to what an oncologist currently provides as "standard of care."
  Arms: Static care plan

SUMMARY:
This study is an NCI-funded, randomized control pilot trial to evaluate: (1) the feasibility and acceptability of a web-based, personalized navigation tool (ConnectedCancerCare) and (2) explore whether the tool improves delivery of team-based survivorship care for women who have recently finished primary breast cancer treatment.

DETAILED DESCRIPTION:
This study is a randomized control pilot trial involving 60 women newly diagnosed with early-stage breast cancer who are finishing primary treatment. Participants will be randomized either to the intervention arm (CCC website that provides information on team-based follow-up care for both cancer surveillance and preventive care) or the control arm (static online survivorship care plan template, adapted from the ASCO breast cancer survivorship template). The feasibility and acceptability of the tool and correlations with patient-reported outcomes will be assessed 3 months following the completion of a baseline survey via an online follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early Stage (0-IIB) breast cancer
* Must be a patient of a University of Michigan Breast Cancer Oncologist
* Must be completing primary cancer treatment and transitioning into survivorship
* Must be able to speak, read and write in English
* Must have access and the ability to use the internet

Exclusion Criteria:

* Diagnosed with stage III or IV breast cancer
* Unable to speak, read, and write in English

Ages: 21 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women being treated at the University of Michigan Rogel Cancer Center for stage 0-2 breast cancer.
Enrollment: 66 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren P Wallner, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 160 eligible women were invited to participate; 66 women enrolled (completed the baseline survey and were randomized).
Groups:
- Control: Static Care Plan: The control arm will receive is a static survivorship care plan template in PDF format that includes information similar to what an oncologist currently provides as "standard of care."
- Intervention: CCC Website: ConnectedCancerCare (CCC) is a web-based guide to support survivorship care for women who have been treated for early-stage (stages 0-II) breast cancer. It encourages patients to utilize team-based care by oncologists and primary care physicians and provides them with the information on cancer surveillance, screenings and preventive healthcare during survivorship.
Period: Overall Study
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Started (Enrolled) | 33 | 33
Completed (Completed the 3-month follow-up survey.) | 26 | 28
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Static Care Plan: The control arm will receive a static survivorship care plan template in PDF format that includes information similar to what an oncologist currently provides as "standard of care."
- CCC Website: ConnectedCancerCare (CCC) is a web- based guide to support survivorship care for women who have been treated for early- stage (stages 0-II) breast cancer. It encourages patients to utilize team-based care by oncologists and primary care physicians and provides them with the information on cancer surveillance, screenings and preventive healthcare during survivorship.
- Total: Total of all reporting groups
Arm/Group | Static Care Plan | CCC Website | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.4) | 57.8 (10.8) | 56.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 29 | 56
  Black | 1 | 1 | 2
  Hispanic | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Other | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  High school/some college | 10 | 13 | 23
  College graduate or more | 23 | 20 | 43
Insurance [Count of Participants; unit: Participants]
  Medicare | 10 | 8 | 18
  Medicaid/Other government | 3 | 1 | 4
  Private | 20 | 24 | 44
Employment [Count of Participants; unit: Participants]
  Employed | 17 | 17 | 34
  Retired | 10 | 8 | 18
  Other not employed | 6 | 8 | 14
Breast Cancer Stage at Diagnosis [Count of Participants; unit: Participants] — Participants self-reported their breast cancer stage at diagnosis, with response options stage 0, stage I, stage II, stage III and stage IV, with higher values representing a higher stage at diagnosis. Population: 11 participants did not self-report this data.
  Participants
    Stage 0: number analyzed (Participants) | 31 | 24 | 55
    Stage 0 | 3 | 2 | 5
    Stage 1: number analyzed (Participants) | 31 | 24 | 55
    Stage 1 | 14 | 15 | 29
    Stage 2: number analyzed (Participants) | 31 | 24 | 55
    Stage 2 | 14 | 7 | 21
Primary Surgical Treatment [Count of Participants; unit: Participants]
  Lumpectomy | 20 | 17 | 37
  Unilateral mastectomy | 5 | 10 | 15
  Bilateral mastectomy | 8 | 6 | 14
Received radiation [Count of Participants; unit: Participants]
  No | 9 | 11 | 20
  Yes | 24 | 22 | 46
Received Chemotherapy [Count of Participants; unit: Participants]
  No | 17 | 19 | 36
  Yes | 16 | 14 | 30
On endocrine therapy [Count of Participants; unit: Participants]
  No | 7 | 2 | 9
  Yes | 26 | 31 | 57
Number of Comorbidities [Count of Participants; unit: Participants]
  0 | 15 | 15 | 30
  1 | 14 | 12 | 26
  2+ | 4 | 6 | 10
Had a primary care provider at enrollment [Count of Participants; unit: Participants]
  No | 2 | 2 | 4
  Yes | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Cancer Patients Successfully Recruited to Participate in the Study
Description: We anticipate a response rate of 80% enrollment (n=60). We will assess the number of patients successfully recruited who enroll and complete the baseline survey.
Time Frame: At baseline survey
Population: Number of eligible women invited to participate
Measure: Count of Participants; unit: Participants
Groups:
- Recruitment Population: Pre-randomization recruitment and enrollment
Arm/Group | Recruitment Population
Number analyzed (Participants) | 160
Participants | 66

2. Secondary Outcome: Rating the Experience With the CCC Web-based, Survivorship Care Plan
Description: Acceptability and usability assessed by the following 6 key factors: 1. Ease of use; 2. Helpful during the transition to survivorship; 3. Helpful in terms of planning when to see my PCP and when to see my Oncologist; 4."Would recommend CCC to other patients"; 5. Length of time it took to go through the website; 6. Amount of information on the website. Each of the 6 factors will be assessed using a 5-point (1-5) Likert scale with higher scores (3, 4, 5) representing better acceptance and usability of the CCC website. Based on prior work, a cut off of 50% or more reporting a score of 3 or higher will be used to measure acceptance within each domain. The average of each participant's responses to the 6 items will result in one score per participant, on a scale of 1 - 5. A single summary score of acceptability across all participants will be determined by averaging the individual scores. On a scale of 1-5, a score of 3 or higher indicates acceptability to the majority of participants.
Time Frame: Follow-Up Survey: 3 months
Population: Intervention arm only; participants who completed the follow-up survey at 3 months post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: CCC Website
Number analyzed (Participants) | 28
score on a scale | 4.4 (2.0)

3. Secondary Outcome: Percentage of Patients Reporting a Preference for an Oncologist vs. PCP for Their Continuing Cancer Care Services
Description: An 8 item list of continuing care services adapted from the CanSORT Provider Roles Scale (iCanCare Study) is used to assess participants' preferences for seeing their Oncologist or PCP.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Control: Static Care Plan: The control arm will receive a static survivorship care plan template in PDF format that includes information similar to what an oncologist currently provides as "standard of care."
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Number analyzed (Participants) | 26 | 28
Participants
  Surveillance (mammogram) | 0 | 3
  Screening for second primary cancers | 5 | 14
  General preventive care | 23 | 25
  Comorbidity management | 24 | 24
  Physical effects | 2 | 3
  Psychological effects | 15 | 20
  Reassurance about recurrence risk | 1 | 1
  Endocrine therapy management | 13 | 15

4. Secondary Outcome: Percentage of Patients Scheduling a Primary Care Physician (PCP) Appointment
Description: The percentage of patients who have scheduled a follow-up visit with their PCP after viewing the CCC web tool (intervention arm) or after receiving the static survivorship care plan (control arm).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Number analyzed (Participants) | 26 | 28
Participants | 11 | 18

5. Secondary Outcome: Patient-Reported Satisfaction With Oncologist/PCP Coordination of Care
Description: A 5-point scale will be used to ask patients to rate their satisfaction with the coordination of care provided by their Oncologist and PCP. The rating scale will range from a value of 1 ('not at all') to a value of 5 ('extremely satisfied'), with a higher numeric value representing greater satisfaction with coordination of care. The mean satisfaction scores will be compared between the intervention and control arms.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Number analyzed (Participants) | 26 | 28
score on a scale | 3.1 (1.2) | 3.7 (1.0)

6. Secondary Outcome: Percentage of Patients That Communicated With PCP About Provider Roles
Description: Communication with PCP about provider roles was measured using an item adapted to the patient perspective from a prior study of providers' views about shared cancer care roles. Patients were asked if they communicated in the past 3 months with their PCP about who will manage specific aspects of their survivorship care (yes/no).
Time Frame: 3 months
Population: Participants who saw a PCP after completing the baseline survey are included in the analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Number analyzed (Participants) | 11 | 18
Participants | 2 | 12

7. Secondary Outcome: Knowledge About Team-based Survivorship Care
Description: Knowledge about team-based survivorship care was measured utilizing an 8-item scale adapted from the Perceived Primary Care Delivery of Survivorship Care Scale. It includes items specific to patients' knowledge of PCPs roles in team-based care delivery, (e.g. second cancer screening, symptom management). The responses were rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The responses to the 8 items were then averaged to create a mean knowledge summary score for each participant, ranging from 1 to 5, with higher values representing greater knowledge about team-based survivorship care.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
Number analyzed (Participants) | 26 | 28
score on a scale | 3.4 (0.9) | 3.7 (0.6)

ADVERSE EVENTS:
Time Frame: Up to 3 months post-enrollment.
Arm/Group | Control: Static Care Plan | Intervention: CCC Website
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03618017/Prot_SAP_001.pdf